CLINICAL TRIAL: NCT03320824
Title: A Randomized, Controlled, Evaluator-Blinded, Multi-Center Study to Evaluate the Effectiveness and Safety of Restylane Kysse Versus a Control in the Augmentation of Soft Tissue Fullness of the Lip
Brief Title: New Dermal Filler for Lip Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USK1701
Record Dates: First submitted 2017-09-27; First posted 2017-10-25 (Actual); Results first posted 2020-06-18 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2020-06

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- New Dermal Filler (Experimental): hyaluronic acid
  Interventions: Device: New Dermal Filler
- Dermal Filler (Active Comparator): hyaluronic acid
  Interventions: Device: Device: FDA Approved Dermal Filler

INTERVENTIONS:
Device: New Dermal Filler — hyaluronic acid
  Arms: New Dermal Filler
Device: Device: FDA Approved Dermal Filler — hyaluronic acid
  Arms: Dermal Filler

SUMMARY:
To demonstrate non-inferiority of Kysse versus a control in lip fullness augmentation

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to comply with the requirements of the study and providing a signed written informed consent.
* Males or non-pregnant, non-breastfeeding females, 22 years of age or older.
* Seeking augmentation therapy for the lips

Exclusion Criteria:

* Allergy of hypersensitivity to any injectable hyaluronic acid gel or to gram positive bacterial proteins.
* Allergy or hypersensitivity to lidocaine or other amide-type anesthetics, or topical anesthetics or nerve blocking agents.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Clinical Testing of Bevelry Hills, Encino, California
  - Cosmetic Laser Dermatology, San Diego, California
  - Art of Skin MD, Solana Beach, California
  - Skin Research Institute, LLC, Coral Gables, Florida
  - University of Miami, Miami, Florida
  - Research Institute of SouthEast, West Palm Beach, Florida
  - Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - Maryland Dermatology, Laser, Skin & Vein Institute, Hunt Valley, Maryland
  - SkinCare Physicians, Chestnut Hill, Massachusetts
  - BOYD, Birmingham, Michigan
  - Laser & Skin Surgery Center of New York, New York, New York
  - Aesthetic Solutions, PA, Chapel Hill, North Carolina
  - Brian S. Biesman, MD, Nashville, Tennessee
  - Center for Advanced Clinical Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Dermal Filler | Dermal Filler
Started | 184 | 89
Completed | 166 | 85
Not Completed | 18 | 4
Not completed — Withdrawal by Subject | 8 | 1
Not completed — Lost to Follow-up | 10 | 1
Not completed — moved out of state | 0 | 1
Not completed — could not complete final visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject randomized to control (Dermal Filler) group but received New Dermal filler in error; therefore they are included in the New Dermal Filler group.Three subjects had baseline MLFS = 5 and were excluded from ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | New Dermal Filler | Dermal Filler | Total
Number analyzed (Participants) | 183 | 87 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (13.5) | 53.6 (10.8) | 52.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 85 | 261
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 15 | 44
  Not Hispanic or Latino | 154 | 72 | 226
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 2 | 9
  White | 173 | 81 | 254
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 183 | 87 | 270
Fitzpatrick Skin Type (FST) [Count of Participants; unit: Participants] — I (White, very fair, red or blond hair, blue eyes, freckles) II (White, fair, red or blond hair; blue, hazel or geen eyes) III (Cream white, fair with any eye or hair color, very common) IV (Brown, typical Mediterranean Caucasian skin) V (Dark brown, Middle Eastern skin type) VI (Black)
  Participants
    FST I | 7 | 4 | 11
    FST II | 77 | 31 | 108
    FST III | 63 | 34 | 97
    FST IV | 23 | 13 | 36
    FST V | 10 | 4 | 14
    FST VI | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Assess Effectiveness of the Treatment Using the Medicis Lip Fullness Scale (MLFS)
Description: The MLFS is a validated photograph-based outcome instrument that is designed specifically for quantifying lip fullness. Scoring of lip fullness (grades 0-5, with a higher score reflecting greater lip fullness) was based on visual live assessment by the Blinded Evaluator at defined time points, and not on a comparison to the baseline appearance. Effectiveness is defined as change from baseline at 8 weeks after last injection of New Dermal Filler or Dermal Filler (control).
Time Frame: 8 weeks after last injection
Measure: Mean (Standard Deviation); unit: Change in MLFS score from baseline
Arm/Group | New Dermal Filler | Dermal Filler
Number analyzed (Participants) | 176 | 85
Change in MLFS score from baseline
  Upper lip | 1.8 (0.96) | 1.7 (0.91)
  Lower lip | 1.8 (0.98) | 1.8 (0.86)

2. Secondary Outcome: Assess Effectiveness of the New Dermal Filler Treatment in the Upper & Lower Lips Using the Medicis Lip Fullness Scale
Description: The MLFS is a validated photograph-based outcome instrument that is designed specifically for quantifying lip fullness. Scoring of lip fullness (grades 0-5, with a higher score reflecting greater lip fullness) was based on visual live assessment by the Blinded Evaluator at defined time points, and not on a comparison to the baseline appearance. Effectiveness is defined as change from baseline at X weeks after last injection of New Dermal Filler.
Time Frame: 16, 24, 32, 40, and 48 weeks after last injection
Population: Observed cases at each visit, New Dermal Filler
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Dermal Filler
Number analyzed (Participants) | 183
score on a scale
  Upper lip Week 16: number analyzed (Participants) | 174
  Upper lip Week 16 | 1.6 (0.92)
  Lower lip Week 16: number analyzed (Participants) | 174
  Lower lip Week 16 | 1.6 (0.96)
  Upper lip Week 24: number analyzed (Participants) | 168
  Upper lip Week 24 | 1.4 (0.94)
  Lower lip Week 24: number analyzed (Participants) | 168
  Lower lip Week 24 | 1.4 (0.98)
  Upper lip Week 32: number analyzed (Participants) | 167
  Upper lip Week 32 | 1.2 (0.91)
  Lower lip Week 32: number analyzed (Participants) | 167
  Lower lip Week 32 | 1.3 (0.94)
  Upper lip Week 40: number analyzed (Participants) | 166
  Upper lip Week 40 | 1.2 (0.98)
  Lower lip Week 40: number analyzed (Participants) | 166
  Lower lip Week 40 | 1.3 (1.00)
  Upper lip Week 48: number analyzed (Participants) | 169
  Upper lip Week 48 | 1.0 (0.91)
  Lower lip Week 48: number analyzed (Participants) | 169
  Lower lip Week 48 | 1.1 (0.94)

3. Secondary Outcome: Assess Effectiveness of the New Dermal Filler Treatment in the Upper & Lower Lips Using the Medicis Lip Fullness Scale
Description: Based on Response Rates (defined as at least 1 point improvement from baseline) after treatment with New Dermal Filler
Time Frame: 16, 24, 32, 40, and 48 weeks
Population: Responder is defined as subjects with at least one point improvement from baseline MLFS (blinded evaluator). Response in both lips concurrently.
Measure: Count of Participants; unit: Participants
Arm/Group | New Dermal Filler
Number analyzed (Participants) | 183
Participants
  Week 16: number analyzed (Participants) | 174
  Week 16 | 142
  Week 24: number analyzed (Participants) | 168
  Week 24 | 129
  Week 32: number analyzed (Participants) | 167
  Week 32 | 115
  Week 40: number analyzed (Participants) | 166
  Week 40 | 110
  Week 48: number analyzed (Participants) | 169
  Week 48 | 101

4. Secondary Outcome: Assess Aesthetic Improvement in the Perioral Rhytids & Oral Commissures After New Dermal Filler Treatment Using the Wrinkle Assessment Scale (Change From Baseline, Blinded Evaluator)
Description: Based on Change from Baseline, New Dermal Filler using WAS. Scoring of the upper perioral rhytids and oral commissures was based on visual live assessment by the Blinded Evaluator at defined time points, and not on a comparison to the baseline appearance. Scoring of fold severity was based on visual assessment of the length and apparent depth of the wrinkle at a certain time-point and measured on a 6-point scale, with 0 being no wrinkle and 5 being very deep wrinkle/redundant fold.
Time Frame: 8, 16, 24, 32, 40, and 48 weeks after last injection
Population: Number observed at each visit, New Dermal Filler
Measure: Mean (Standard Deviation); unit: change in WAS score from baseline
Arm/Group | New Dermal Filler
Number analyzed (Participants) | 183
change in WAS score from baseline
  Upper Perioral Lines, Week 8: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 8 | -2.2 (0.99)
  Upper Perioral Lines, Week 16: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 16 | -1.8 (0.97)
  Upper Perioral Lines, Week 24: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 24 | -1.7 (0.95)
  Upper Perioral Lines, Week 32: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 32 | -1.6 (1.00)
  Upper Perioral Lines, Week 40: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 40 | -1.5 (0.87)
  Upper Perioral Lines, Week 48: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 48 | -1.6 (1.04)
  Left oral commissure Week 8: number analyzed (Participants) | 134
  Left oral commissure Week 8 | -1.5 (1.11)
  Right oral commissure Week 8: number analyzed (Participants) | 133
  Right oral commissure Week 8 | -1.4 (1.05)
  Left oral commissure Week 16: number analyzed (Participants) | 132
  Left oral commissure Week 16 | -1.4 (1.19)
  Right oral commissure Week 16: number analyzed (Participants) | 131
  Right oral commissure Week 16 | -1.3 (1.08)
  Left oral commissure Week 24: number analyzed (Participants) | 130
  Left oral commissure Week 24 | -1.3 (1.05)
  Right oral commissure Week 24: number analyzed (Participants) | 129
  Right oral commissure Week 24 | -1.2 (1.11)
  Left oral commissure Week 32: number analyzed (Participants) | 129
  Left oral commissure Week 32 | -1.3 (1.24)
  Right oral commissure Week 32: number analyzed (Participants) | 128
  Right oral commissure Week 32 | -1.2 (1.14)
  Left oral commissure Week 40: number analyzed (Participants) | 130
  Left oral commissure Week 40 | -1.1 (1.30)
  Right oral commissure Week 40: number analyzed (Participants) | 129
  Right oral commissure Week 40 | -1.1 (1.21)
  Left oral commissure Week 48: number analyzed (Participants) | 131
  Left oral commissure Week 48 | -1.2 (1.28)
  Right oral commissure Week 48: number analyzed (Participants) | 130
  Right oral commissure Week 48 | -1.1 (1.25)

5. Secondary Outcome: Assess Aesthetic Improvement in the Perioral Rhytids & Oral Commissures After New Dermal Filler Treatment Using the Wrinkle Assessment Scale (Response Rates, Blinded Evaluator)
Description: Based on Response Rates (defined as at least 1 point improvement from baseline), New Dermal Filler using WAS. Scoring of the upper perioral rhytids and oral commissures was based on visual live assessment by the Blinded Evaluator at defined time points, and not on a comparison to the baseline appearance. Scoring of fold severity was based on visual assessment of the length and apparent depth of the wrinkle at a certain time-point and measured on a 6-point scale, with 0 being no wrinkle and 5 being very deep wrinkle/redundant fold. .
Time Frame: 8, 16, 24, 32, 40, and 48 weeks
Population: Observed cases at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | New Dermal Filler
Number analyzed (Participants) | 183
Participants
  Upper Perioral Lines, Week 8: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 8 | 50
  Upper Perioral Lines, Week 16: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 16 | 47
  Upper Perioral Lines, Week 24: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 24 | 47
  Upper Perioral Lines, Week 32: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 32 | 47
  Upper Perioral Lines, Week 40: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 40 | 47
  Upper Perioral Lines, Week 48: number analyzed (Participants) | 53
  Upper Perioral Lines, Week 48 | 44
  Left oral commissure Week 8: number analyzed (Participants) | 134
  Left oral commissure Week 8 | 106
  Left oral commissure Week 16: number analyzed (Participants) | 132
  Left oral commissure Week 16 | 102
  Left oral commissure Week 24: number analyzed (Participants) | 130
  Left oral commissure Week 24 | 98
  Left oral commissure Week 32: number analyzed (Participants) | 129
  Left oral commissure Week 32 | 94
  Left oral commissure Week 40: number analyzed (Participants) | 130
  Left oral commissure Week 40 | 87
  Left oral commissure Week 48: number analyzed (Participants) | 131
  Left oral commissure Week 48 | 90
  Right oral commissure Week 8: number analyzed (Participants) | 133
  Right oral commissure Week 8 | 104
  Right oral commissure Week 16: number analyzed (Participants) | 131
  Right oral commissure Week 16 | 101
  Right oral commissure Week 24: number analyzed (Participants) | 129
  Right oral commissure Week 24 | 97
  Right oral commissure Week 32: number analyzed (Participants) | 128
  Right oral commissure Week 32 | 89
  Right oral commissure Week 40: number analyzed (Participants) | 129
  Right oral commissure Week 40 | 86
  Right oral commissure Week 48: number analyzed (Participants) | 130
  Right oral commissure Week 48 | 83

6. Secondary Outcome: Assess Overall Aesthetic Improvement After New Dermal Filler Treatment Using the Global Aesthetic Improvement Scale Determined by Response Rates, Subject Assessment
Description: Responders defined as at least "improved" (improved, much improved, very much improved) as assessed by subject, upper and lower lip combined, New Dermal Filler
Time Frame: 8, 16, 24, 32, 40, and 48 weeks
Population: Observed cases at each visit, New Dermal Filler
Measure: Count of Participants; unit: Participants
Arm/Group | New Dermal Filler
Number analyzed (Participants) | 183
Participants
  Week 8: number analyzed (Participants) | 178
  Week 8 | 170
  Week 16: number analyzed (Participants) | 175
  Week 16 | 161
  Week 24: number analyzed (Participants) | 169
  Week 24 | 148
  Week 32: number analyzed (Participants) | 167
  Week 32 | 140
  Week 40: number analyzed (Participants) | 167
  Week 40 | 131
  Week 48: number analyzed (Participants) | 169
  Week 48 | 132

7. Secondary Outcome: Assess Overall Aesthetic Improvement After New Dermal Filler Treatment Using the Global Aesthetic Improvement Scale, Treating Investigator
Description: Determined by Response Rates, Treating Investigator Assessment, New Dermal Filler
Time Frame: 8, 16, 24, 32, 40, and 48 weeks
Population: Observed cases at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | New Dermal Filler
Number analyzed (Participants) | 183
Participants
  Upper and lower lip combined, Week 8: number analyzed (Participants) | 178
  Upper and lower lip combined, Week 8 | 175
  Upper and lower lip combined, Week 16: number analyzed (Participants) | 175
  Upper and lower lip combined, Week 16 | 169
  Upper and lower lip combined, Week 24: number analyzed (Participants) | 168
  Upper and lower lip combined, Week 24 | 145
  Upper and lower lip combined, Week 32: number analyzed (Participants) | 167
  Upper and lower lip combined, Week 32 | 137
  Upper and lower lip combined, Week 40: number analyzed (Participants) | 167
  Upper and lower lip combined, Week 40 | 121
  Upper and lower lip combined, Week 48: number analyzed (Participants) | 169
  Upper and lower lip combined, Week 48 | 114

8. Secondary Outcome: Assessment of Improvement in Lip Fullness After New Dermal Filler Treatment, by Independent Photographic Reviewer
Description: Proportion of Improvement (Responders) Based on Independent Photographic Reviewer Assessment by Weeks after Last Injection, New Dermal Filler
Time Frame: 8, 24, 40, and 48 weeks
Population: Observed cases at each visit. Response is defined as an improvement from baseline assessed via random, blinded pairing and review of the baseline and post-baseline photographs
Measure: Count of Participants; unit: Participants
Arm/Group | New Dermal Filler
Number analyzed (Participants) | 183
Participants
  Upper lip, Week 8: number analyzed (Participants) | 172
  Upper lip, Week 8 | 168
  Lower lip, Week 8: number analyzed (Participants) | 172
  Lower lip, Week 8 | 164
  Upper lip, Week 24: number analyzed (Participants) | 163
  Upper lip, Week 24 | 149
  Lower lip, Week 24: number analyzed (Participants) | 163
  Lower lip, Week 24 | 144
  Upper lip, Week 40: number analyzed (Participants) | 164
  Upper lip, Week 40 | 149
  Lower lip, Week 40: number analyzed (Participants) | 164
  Lower lip, Week 40 | 138
  Upper lip, Week 48: number analyzed (Participants) | 167
  Upper lip, Week 48 | 152
  Lower lip, Week 48: number analyzed (Participants) | 167
  Lower lip, Week 48 | 147

9. Secondary Outcome: Assess Subject Satisfaction With New Dermal Filler Treatment Using the FACE-Q
Description: Subjects' satisfaction using the validated FACE-Q scales Satisfaction with Lips and Appraisal of Lines: Lips at baseline and at Week 8, 16, 24, 32, 40, and 48 weeks after last injection based on individual questions in each questionnaire as well as the Rasch transformed total scores and the change from baseline in the Rasch transformed scores. Rasch-transformed total score (0-100) according the FACE-Q manual; the higher total score indicated greater subject satisfaction.A positive change from baseline indicates an improvement. Baseline is defined as the last observation before initial treatment takes place at the baseline visit on Day 1.
Time Frame: 8, 16, 24, 32, 40, and 48 weeks
Population: Observed cases at each visit, New Dermal Filler
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Dermal Filler
Number analyzed (Participants) | 183
score on a scale
  Baseline | 28.1 (16.47)
  Week 8: number analyzed (Participants) | 177
  Week 8 | 83.3 (20.23)
  Week 16: number analyzed (Participants) | 175
  Week 16 | 76.2 (24.06)
  Week 24: number analyzed (Participants) | 169
  Week 24 | 74.9 (24.34)
  Week 32: number analyzed (Participants) | 167
  Week 32 | 72.0 (24.02)
  Week 40: number analyzed (Participants) | 167
  Week 40 | 69.0 (25.48)
  Week 48: number analyzed (Participants) | 169
  Week 48 | 66.3 (26.68)

10. Other Pre Specified Outcome: Evaluate All Reported Adverse Events
Time Frame: 48 weeks
Population: Safety population, Initial and Touch-up Treatment. One subject randomized to the dermal filler group received the new dermal filler in error. This subject is included in the new dermal filler group for safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | New Dermal Filler | Dermal Filler
Number analyzed (Participants) | 185 | 88
Participants
  Treatment Emergent Adverse Event (TEAE) | 72 | 31
  Serious TEAE | 2 | 0
  TEAE related to product and/or injection procedure | 39 | 22
  Serious TEAEs, related | 0 | 0
  Unrelated TEAE | 44 | 22
  No TEAEs | 113 | 57

ADVERSE EVENTS:
Time Frame: 1 year
Description: One subject randomized to the dermal filler group received the new dermal filler in error. This subject is included in the new dermal filler group for safety analysis.
Arm/Group | New Dermal Filler | Dermal Filler
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/88
Serious Adverse Events (participants affected / at risk) | 2/185 | 0/88
Other Adverse Events (participants affected / at risk) | 43/185 | 25/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Dermal Filler (N=185) | Dermal Filler (N=88)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Dermal Filler (N=185) | Dermal Filler (N=88)
Injection site bruising (General disorders) | 14 (37) | 9 (71) — Related
injection site mass (General disorders) | 19 (34) | 10 (22) — Related
injection site nodule (General disorders) | 10 (18) | 6 (18) — Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree not to present or publish any data or reports collected individually or by subgroup of sites prior to full, initial publication based on all data obtained from all sites.

DOCUMENTS (2):
  • Study Protocol (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT03320824/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03320824/SAP_003.pdf